CLINICAL TRIAL: NCT02228291
Title: The Effect of Citric Flavonoid Administration on Endothelial Function and Gut Barrier Function
Brief Title: The Effect of Citric Flavonoid on Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Bouke Salden, Coordinating Investigator, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-3-019
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Obesity; Overweight
Keywords: Polyphenols; Endothelial function; Gut barrier function
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Cellulose
  Interventions: Dietary Supplement: Placebo
- Citric flavonoid (Experimental): Citric flavonoid
  Interventions: Dietary Supplement: Capsule containing citrus flavonoid

INTERVENTIONS:
Dietary Supplement: Capsule containing citrus flavonoid
  Arms: Citric flavonoid
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel study aims to determine the 6-week and acute effects of daily administration of a citrus flavonoid on cardiovascular and intestinal health as assessed by investigation of endothelial function, blood pressure and heart rate, glucose/insulin metabolism, lipid profile and gut barrier function in overweigh subjects.

Futhermore we aim to relate the specific intestinal (microbial) metabolism with final serum levels of specific metabolites of the study product.

ELIGIBILITY:
Inclusion Criteria:

* Overweight men/women (BMI 25-35 kg/m2)
* Healthy individuals
* Age between 18 and 70 years
* Fasting glucose < 7.0 mmol/L
* Normal HbA1c (4.4 to 6.2%)

Exclusion Criteria:

* Type 2 diabetes mellitus (defined as fasting plasma glucose ≥ 7.0 mmol/L)
* Gastroenterological diseases or abdominal surgery
* Cardiovascular diseases, cancer, liver or kidney malfunction, thyroid disorders, disease with a life expectancy shorter than 5 years
* Self-admitted HIV-positive status
* Abuse of products; alcohol (> 20 alcoholic consumptions per week) and drugs
* Smoking
* Plans to lose weight or following a hypocaloric diet during the study period
* Weight gain or loss > 3 kg in previous 3 months
* Use of medication interfering with endpoints
* Intake of antihypertensive medication, statins, corticosteroids, NSAIDs, ciclosporin A, rifampicin are strictly forbidden
* Use of antioxidants, minerals and vitamin supplements available in pharmacies, drugstores, food markets or in alternative medicine
* Hormone replacement therapy (women)
* Use of antibiotics in the 90 days prior to the start of study
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator) in the 180 days prior to the study
* Known pregnancy (assessed by a pregnancy test before start of study), lactation
* Blood donation within 3 months before study period
* Failure to comply prohibited intake of hesperidin containing food products during study period and prohibited intake of food products that are able to influence the FMD measurements one day prior to test days.
* History of any side effects towards the intake of flavonoids or citrus fruits

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 6 weeks
  The primary objective of this study is to evaluate the efficacy on endothelial function, as assessed by flow mediated dilatation (FMD) measurements, after 6 weeks of administration of study product.

SECONDARY OUTCOMES:
Endothelial function | 6 weeks
  The second secondary objective of this study is to determine the 6-week effect on plasma biomarkers of endothelial dysfunction and low-grade inflammation.
Blood pressure & heart rate | 6 weeks
  The third objective of this study is to assess the 6-week effect on blood pressure and heart rate by measuring systolic and diastolic blood pressure and heart rate.
Glucose / insulin metabolism | 6 weeks
  The fourth secondary objective of this study is to determine the 6-week effect on glucose / insulin metabolism by blood measurements.
Lipid profile | 6 weeks
  The fourth secondary objective of this study is to determine the 6-week effect on lipid profile by blood measurements.
Gut barrier function | 6 weeks
  The fifth secondary objective of this study is to assess the acute and 6-week effect on gut barrier function by measuring plasma and fecal endotoxin (LPS) and zonulin.
Gut barrier function | 6 weeks
  The sixth secondary objective of this study is to assess the 6-week effect of on gut barrier function by performing a gut sugar permeability test.
Colonic inflammation | 6 weeks
  The seventh secondary objective of this study is to assess the 6-week effect on colonic inflammation, by measuring fecal calprotectin.
Bioavailability and metabolism | 5 days
  The eight secondary objective of this study is to enlarge the understanding of the bioavailability and metabolism of this study product in human beings, by relating specific intestinal (microbial) metabolism with serum levels of its metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: A.A.M. Masclee, MD, PhD, Principal Investigator — Department of Internal Medicine, Division of Gastroenterology-Hepatology
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Salden BN, Troost FJ, de Groot E, Stevens YR, Garces-Rimon M, Possemiers S, Winkens B, Masclee AA. Randomized clinical trial on the efficacy of hesperidin 2S on validated cardiovascular biomarkers in healthy overweight individuals. Am J Clin Nutr. 2016 Dec;104(6):1523-1533. doi: 10.3945/ajcn.116.136960. Epub 2016 Oct 26. PMID 27797708